CLINICAL TRIAL: NCT00315458
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Determine Efficacy and Safety of Buprenorphine Transdermal System in Subjects With Moderate To Severe Osteoarthritis Pain Requiring Daily Treatment With Opioids
Brief Title: Buprenorphine Transdermal Patch in Subjects With Osteoarthritis Pain Requiring Opioids. Includes a 52-Week Safety Extension.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP3011 and BUP3011S; NCT01137279 (obsolete NCT alias)
Record Dates: First submitted 2006-04-17; First posted 2006-04-18 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; opioid; transdermal
MeSH Terms: conditions — Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BTDS (Experimental): Buprenorphine transdermal patches 10 or 20 mcg/h
  Interventions: Drug: Buprenorphine transdermal patch
- Placebo (Placebo Comparator): Placebo to match buprenorphine transdermal patch 10 or 20
  Interventions: Drug: Placebo transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch applied for 7-day wear.
  Other Names: Butrans™
  Arms: BTDS
Drug: Placebo transdermal patch — Placebo to match buprenorphine transdermal patch 10 or 20.
  Arms: Placebo

SUMMARY:
The original objective of this study was to assess the safety and efficacy of the buprenorphine transdermal system (BTDS) (5, 10, and 20) in comparison to placebo transdermal system in subjects with moderate to severe osteoarthritis pain. However, this study was terminated early with only 35% of the planned sample size, therefore the primary objective is changed to focus on the safety evaluations.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* clinical evidence of osteoarthritis of the hip, knee, or spine joint for ≥ 1 year currently adequately treated with short acting opioids.
* taking ≥ 30 and ≤ 80 mg oral morphine or morphine equivalents per day for ≥ 2 weeks for control of their osteoarthritis pain.

Exclusion Criteria:

* requiring frequent analgesic therapy for chronic condition(s), other than osteoarthritis of the hip, knee, or spine.
* scheduled for surgery of the disease site (e.g., major joint replacement surgery), or any other major surgery that would fall within the study period.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Parkway Medical Center, Birmingham, Alabama
  - Clinical Research Consultants, Birmingham, Alabama
  - Winston Physician Services, Inc, Haleyville, Alabama
  - Private Practice, Muscle Shoals, Alabama
  - Clinic for Rheumatic Diseases, Tuscaloosa, Alabama
  - Radiant Research, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - ACRC/Arizona Clinical Research, Tuscon, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southbay Pharma Research, Buena Park, California
  - Torrence Clinical Research, Torrance, California
  - Comprehensive Neuroscience Inc, Boynton Beach, Florida
  - Chiefland Medical Center, Chiefland, Florida
  - University Clinical Research Deland, DeLand, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - Drug Study Institute, Jupiter, Florida
  - Coastal Medical Research, Orange City, Florida
  - Ormond Medical Arts Pharmaceutical Res Ctr, Ormond Beach, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Avancia Research, Pembroke Pines, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gold Coast Research LLC, Weston, Florida
  - Georgia Medical Research Institute, Marietta, Georgia
  - Internal Medicine Northwest, Gurnee, Illinois
  - MediSphere Medical Research Center, Evansville, Indiana
  - University of Louisville Medical/Rheumatology, Louisville, Kentucky
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Future Care Studies, Springfield, Massachusetts
  - Bay Area Health Clinic, Bay City, Michigan
  - Medex Healthcare Research Inc, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Health Research Institute, Oklahoma City, Oklahoma
  - Keystone Clinical Solutions, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - BioMedical Research Associates, Shippensburg, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Low Country Rheumatology, Charleston, South Carolina
  - Brown Clinic, Watertown, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - CSS Research, Memphis, Tennessee
  - Prime Care Medical Center, Selmer, Tennessee
  - Team Research of Central Texas, Harker Heights, Texas
  - Quality Research, San Antonio, Texas
  - Advanced Pain Management and Rehab Hilltop Med Center, Virginia Beach, Virginia
  - Sentara Medical Group, Virginia Beach, Virginia
  - Physicians Clinic of Spokane, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12-Dec-2003 (First Patient First Visit) 02-Mar-2005 (Last Patient Last Visit of Extension). At the time of early termination, 39 centers had screened subjects, 22 centers had randomized subjects to the double-blind phase.
Pre-assignment Details: All subjects (N = 159) in the run-in period received BTDS 5 for the first 3 days, titrated to BTDS 10 or 20, continued stable nonopioid analgesic regimen for osteoarthritis (OA) pain, and took oxycodone immediate-release 5-mg capsules as supplemental analgesic therapy for primary OA pain site. N = 107 completed the run-in and were randomized.
Groups:
- Double-blind Placebo Patch: Reference Treatment placebo 10 or 20 applied for 7-day wear
- Double-blind BTDS 10/20: Test treatments buprenorphine transdermal patch (BTDS) 10 or BTDS 20 applied for 7-day wear
- Run-in Period BTDS 5/10/20: All subjects were started on BTDS 5 and titrated to BTDS 10 and 20. Subjects who met the protocol-specified criteria for adequate analgesia were eligible for entry into the double-blind phase. Subjects who could not tolerate at least BTDS 10 were discontinued from the study.
- Extension Phase BTDS 5/10/20: Subjects who finished the entire 12-week (84-day) double-blind phase were eligible to participate in the open-label extension phase. Subjects began treatment with BTDS 5 and their doses were titrated to BTDS 10 or BTDS 20 as needed.
Period: Overall Study
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS 10/20 | Run-in Period BTDS 5/10/20 | Extension Phase BTDS 5/10/20
Started | 51 | 56 | 159 | 39
Completed | 48 | 44 | 107 | 10
Not Completed | 3 | 12 | 52 | 29
Not completed — Administrative | 0 | 3 | 8 | 21
Not completed — Adverse Event | 2 | 4 | 23 | 3
Not completed — Lost to Follow-up | 1 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 20 | 1
Not completed — Did not qualify | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Double-blind BTDS: Test treatments buprenorphine transdermal patch (BTDS) 10 or BTDS 20 applied for 7-day wear
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS | Total
Number analyzed (Participants) | 51 | 56 | 107
Age Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.36) | 59.4 (9.56) | 60.3 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety
Description: For the Run-in and double-blind phases of the study, the focus of this study was changed before unblinding to a safety study due to early termination and having enrolled only 35% of the planned sample size. Therefore, the safety data is presented for the run-in and double-blind and overall exposure to BTDS, which includes the extension phase.
Time Frame: 483 days
Population: The full analysis population consisted of all subjects who were randomized into the double-blind phase and received at least 1 dose of double-blind treatment.
Measure: Number; unit: participants
Groups:
- Double-blind Placebo: Reference treatment placebo 10 or 20 applied for 7-day wear
- Double-blind BTDS: Test treatment buprenoprhine transdermal patch (BTDS) 10 or BTDS 20 applied for 7-day wear
- Run-in Period: All subjects were started on BTDS 5 and titrated to BTDS 10 and 20. Subjects who met the protocol-specified criteria for adequate analgesia were eligible for entry into the double-blind phase. Subjects who could not tolerate at least BTDS 10 were discontinued from the study.
- Overall BTDS Exposure: Total number of subjects exposed to BTDS for overall study which includes the core study and extension phase.
Arm/Group | Double-blind Placebo | Double-blind BTDS | Run-in Period | Overall BTDS Exposure
Number analyzed (Participants) | 51 | 56 | 159 | 159
participants
  Death | 0 | 1 | 0 | 1
  Serious adverse events | 1 | 2 | 1 | 5
  All Other Adverse Events in ≥ 4.5% of Subjects | 14 | 22 | 60 | 82

ADVERSE EVENTS:
Time Frame: Subjects with AEs that were ongoing at subject's last study visit were followed until resolution or 30 days after last visit, whichever came first. AEs reported during 7 days following last visit were followed until resoultion or 30 days after last visit.
Description: AEs were learned of through spontaneous reports and subject interview.
Groups:
- Double-blind BTDS 10/20: Test treatment buprenorphine transdermal patch (BTDS) 10 or BTDS 20 applied for 7-day wear
- Run-in Period: Open-label Run-in period (BTDS 5, 10, or 20) applied for 7-day wear
Arm/Group | Double-blind Placebo Patch | Double-blind BTDS 10/20 | Run-in Period | Overall BTDS Exposure
Serious Adverse Events (participants affected / at risk) | 1/51 | 2/56 | 1/159 | 5/159
Other Adverse Events (participants affected / at risk) | 14/51 | 22/56 | 60/159 | 82/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo Patch (N=51) | Double-blind BTDS 10/20 (N=56) | Run-in Period (N=159) | Overall BTDS Exposure (N=159)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Acute myocardial infarction - DEATH (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — DEATH (systematic and nonsystematic assessments)
Cervical spinal stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Acute exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Systematic and nonsystematic assessments
Recurrent Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Near Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessments
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Systematic and non-systematic assessments.
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Placebo Patch (N=51) | Double-blind BTDS 10/20 (N=56) | Run-in Period (N=159) | Overall BTDS Exposure (N=159)
Nausea (Gastrointestinal disorders) | 4 | 6 | 25 | 32 — Systematic and nonsystematic assessment
Constipation (Gastrointestinal disorders) | 0 | 4 | 10 | 15 — Systematic and nonsystematic assessment
Application site pruritus (General disorders) | 6 | 7 | 16 | 23 — Systematic and nonsystematic assessment
Application site erythema (General disorders) | 3 | 2 | 6 | 9 — Systematic and nonsystematic assessment
Application site rash (General disorders) | 0 | 6 | 1 | 8 — Systematic and nonsystematic assessment
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 5 — Systematic and nonsystematic assessment
Headache (Nervous system disorders) | 5 | 2 | 16 | 22 — Systematic and nonsystematic assessment
Sweating Increased (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 (1) | 6 — Systematic and nonsystematic assessment
Somnolence (Nervous system disorders) | 1 | 0 | 11 | 12 — Systematic and nonsystematic assessment
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 8 — Systematic and nonsystematic assessment
Dizziness (Nervous system disorders) | 0 | 2 | 6 | 11 — Systematic and nonsystematic assessment

LIMITATIONS AND CAVEATS:
This study was terminated early for administrative reasons. The efficacy data are not presented since the primary objective of this study was changed identifying it as a safety study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days